CLINICAL TRIAL: NCT00971152
Title: Effect of a Higher Than Maximum 450IU Gonadotropin Dose on Patient Outcomes in an In-Vitro Fertilization Setting: a Randomized Controlled Non-infertility Trial
Brief Title: Effect of a Higher Than Maximum 450IU Gonadotropin Dose in an In-vitro Fertilization Cycle
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Clinique Ovo (Industry)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F-GYN-08-02
Record Dates: First submitted 2009-09-02; First posted 2009-09-03 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Subfertility
Keywords: IVF; dose comparison of gonadotrophins; poor responder to ovarian stimulation
MeSH Terms: conditions — Infertility | interventions — Menotropins; Injections; Urofollitropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 450 IU daily dose of gonadotrophin (Active Comparator)
  Interventions: Drug: menotropins for injection; Drug: urofollitropin for injection
- 600 IU daily dose of gonadotrophin (Experimental)
  Interventions: Drug: menotropins for injection; Drug: urofollitropin for injection

INTERVENTIONS:
Drug: menotropins for injection — comparison of different dosages
  Other Names: Menopur
Drug: urofollitropin for injection — comparison of different dosages
  Other Names: Bravelle

SUMMARY:
This goal of this study is to evaluate the outcomes from in vitro fertilization cycles where a 450 IU daily dose of gonadotropins is administered compared to those where a 600 IU daily dose is administered for women who are at risk of a poor ovarian response in order to determine if one dose or the other results in improved cycle outcomes.

ELIGIBILITY:
Inclusion Criteria:

* RESIDENT OF CANADA
* Premenopausal
* Age 40 years or less at the time of enrollment
* At risk of a poor ovarian response defined as: either <5 oocytes or <8 follicles in a previous cycle, FSH > 10 IU/L, AMH < 1 pg/ml , antral follicle count less or equal to 8 or previous IVF cancellation
* Primary infertility or secondary
* Not previously undertaken a cycle that was included in this study

Exclusion Criteria:

* Simultaneous participation in another clinical trial
* Body mass index (BMI) > 38 kg/m2
* Early follicular phase (day 2-4) serum FSH level > 20 mIU/ml
* Any contraindication to being pregnant and carrying a pregnancy to term
* Contraindication for the use of Estrace® , Suprefact®, Menopur®, Bravelle®, hCG, and luteal phase support medication
* Any ovarian or abdominal abnormality that may interfere with adequate transvaginal ultrasound evaluation
* Administration of any investigational drugs within three months prior to study enrollment
* Patient not able to communicate adequately with the investigators and to comply with the requirements of the entire study
* Positive results of screening of either partner for HIV antibodies, Hepatitis B (other than for surface antibodies present after vaccination) or Hepatitis C
* Unwillingness to give written informed consent

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 366 (Actual)
Dates: Start 2009-09; Primary Completion 2013-10 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Number of metaphase II oocytes retrieved during the course of one treatment cycle | 2 years

SECONDARY OUTCOMES:
Number of follicles recruited per patient during stimulation | 2 years
Fertilization rate per patient (number of normally fertilized (with 2 pronuclei) oocytes/number of mature oocytes collected) | 2 years
Embryo cleavage rate per patient (number of divided normally fertilized oocytes/number of normally fertilized oocytes) | 2 years
Number of embryos available per patient | 2 years
Number of supernumerary embryos available for cryopreservation per patient | 2 years
Implantation rate | 2 years
Biochemical pregnancy rate | 2 years
Clinical pregnancy rate | 2 years
Rate of multiple gestation | 2 years
Ongoing pregnancy rate | 2 years
Live birth rate | 2 years
rate of occurrence of ovarian hyperstimulation syndrome (OHSS) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Louise Lapensee, MD, Principal Investigator — ovo fertilité; Jacques Kadoch, MD, Study Director — OVO Fertilité and OVO R & D
Locations (1):
- Ovo Fertilité, Montreal, Quebec, Canada

REFERENCES:
- [Background] Srouji SS, Missmer SA, Ginsburg ES (2004) Impact of increasing gonadotropins > 450 IU on cycle outcome. Brigham and Women's Hospital, Boston, MA. Fertil Steril 82 (Suppl 2): P292.
- [Background] Flisser E, Krey LC, Berkeley AS (2005) Diminishing Returns of Increasing Gonadotropin Dosage in Subsequent In Vitro Fertilization (IVF) Cycles?. Fertil Steril 84 (Suppl 1) P483.
- [Derived] Lefebvre J, Antaki R, Kadoch IJ, Dean NL, Sylvestre C, Bissonnette F, Benoit J, Menard S, Lapensee L. 450 IU versus 600 IU gonadotropin for controlled ovarian stimulation in poor responders: a randomized controlled trial. Fertil Steril. 2015 Dec;104(6):1419-25. doi: 10.1016/j.fertnstert.2015.08.014. Epub 2015 Sep 8. PMID 26361207
- See also: OVO fertilité website — http://www.ovoclinic.com/